CLINICAL TRIAL: NCT01884649
Title: Fetuin A as a New Marker of Inflammation in Hashimoto Thyroiditis
Brief Title: Fetuin A in Hashimoto Thyroiditis
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Sevilay Muratli, M.D., Istanbul Medeniyet University
Other Study IDs: GEAH-1
Record Dates: First submitted 2013-06-17; First posted 2013-06-24 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Hashimoto Thyroiditis
Keywords: Acute phase reactant, fetuin A, Hashimoto thyroiditis
MeSH Terms: conditions — Hashimoto Disease

STUDY DESIGN:
Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group of Hashimoto thyroiditis patients
- Healty control group

SUMMARY:
Fetuin-A levels are reported to be low as a negative acute phase reactant in systemical inflammatory situations. Hashimoto thyroiditis is characterized with inflammation. In this study, we hypothesised that the serum fetuin A levels could be found to be low due to inflammation in patients with Hashimoto thyroiditis

DETAILED DESCRIPTION:
Patients ≥ 20 years of age being followed up at the outpatient clinics of the Internal Medicine Department in Medeniyet University Goztepe Training and Research Hospital and fulfilling the eligibility criteria will be included in the study. Approval of the local ethics committee and informed consent of the participants will be received for the study. The study is conducted in accordance with the Declaration of Helsinki. Demographic characteristics, concomitant diseases, smoking and alcohol drinking habits, concomitant medication usage, anthropometric and biochemistry data of the eligible patients will be recorded. Patient group will consist of patients with newly diagnosed Hashimoto thyroiditis and the control group will consist of healthy volunteers.

Groups will be compared according to their demographic, an¬thropometric and biochemistry data and serum fetuin-A levels. In order to detect the relationship between the serum fetuin-A levels and clinical features, correlation analyses will be done.

ELIGIBILITY:
Inclusion Criteria:

* patients newly diagnosed with Hashimoto thyroiditis

Exclusion Criteria:

* Acute infection
* Acute or chronic inflammatory disease
* Anti-inflammatory treatment (non-steroidal anti-inflammatory, corticosteroids etc.)
* Hypoxic situations (chronic obstructive pulmonary disease etc.)
* Severe heart, kidney and liver disease
* Pregnancy
* Endocrine disorders
* Malignancy
* Usage of drug that affects thyroid hormone levels

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 20 years of age being followed up at the outpatient clinics of the Internal Medicine Department in Medeniyet University Goztepe Training and Research Hospital and fulfilling the below mentioned criteria were included in the study
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Comparison of serum fetuin A levels between patients with Hashimoto thyroiditis and healthy subjects | 1 day (The blood samples were obtained on the same day participants arrived to outpatient clinics.)